CLINICAL TRIAL: NCT00004799
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Acellular and Whole-Cell Pertussis Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Bacteriological Laboratory (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 199/11953; NBL-SS-19910415
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-01

CONDITIONS: Pertussis
Keywords: bacterial infection; immunologic disorders and infectious disorders; pertussis; rare disease
MeSH Terms: conditions — Whooping Cough; Bacterial Infections; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Diphtheria-Tetanus Vaccine

INTERVENTIONS:
Biological: whole-cell pertussis vaccine
Biological: diphtheria-tetanus vaccine

SUMMARY:
OBJECTIVES: I. Compare the safety and efficacy of acellular 2-component vs. acellular multicomponent vs. whole-cell pertussis vaccine vs. placebo in infants living in Sweden.

II. Compare the relative protection of each vaccine against atypical or subclinical pertussis infection.

III. Analyze possible laboratory correlates to vaccine protection.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution.

The first group of infants receives a vaccine composed of inactivated pertussis toxin (iPT) and filamentous hemagglutin (FHA).

The second group receives a vaccine containing iPT, FHA, pertactin, agglutinogen 2, and agglutinogen 3.

The third group receives a whole-cell pertussis vaccine. The fourth group receives a diphtheria-tetanus vaccine as the control. All vaccines are given as an intramuscular injection, at 2-3, 4, and 6 months of age.

Close surveillance of infants and families continues for 2-3 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Population Characteristics--

* Infants aged 2 months at planned date of first vaccination
* No prior pertussis confirmed by culture
* The following do not exclude: Down syndrome Prematurity Healthy babies vaccinated according to chronological age Recent pertussis exposure Seizures in parent or sibling Sudden infant death in sibling Close relative with history of anaphylaxis or allergy Close relative with history of strong reaction to vaccination

--Patient Characteristics--

* Age: Under 3 months
* Renal: No renal failure
* Other: No prior gammaglobulin No requirement for immunosuppressives, e.g., HIV infection No manifest immunosuppression No serious chronic illness associated with failure to thrive No cardiac disease No progressive neurologic disease No uncontrolled epilepsy or infantile spasms No parental language or communication barrier

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10000
Dates: Start 1991-04

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Olin, Study Chair — National Bacteriological Laboratory